CLINICAL TRIAL: NCT04186533
Title: A Default Option for Health: Improving Nutrition Within the Financial and Geographic Constraints of Food Insecurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Albany (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Julia Hormes, Associate Professor, University at Albany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-E-224-01
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Food Selection; Obesity
Keywords: food insecurity; nutrition; obesity; default option; online grocery shopping
MeSH Terms: conditions — Food Preferences; Obesity | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Default Intervention (Experimental): Participants in the default condition were presented with a pre-filled online shopping cart containing a combination of groceries that meet macro- and micronutrient requirements for their gender and age, and told that they are free to delete, add, and exchange any item they wish to finalize their selections.
  Interventions: Behavioral: Default Option
- Nutrition Education (Active Comparator): Participants in the nutrition education condition were instructed to read brief nutrition education handouts before online grocery shopping.
  Interventions: Behavioral: Nutrition Education

INTERVENTIONS:
Behavioral: Default Option — The default option is a behavioral economics construct that refers to the option a consumer selects if no active choice is made (e.g. opt-out 401K plans, which significantly increase enrollment, compared to active sign up). Participants in the default condition were presented with a prefilled online shopping cart containing groceries that met nutritional requirements based on participants' gender and age.
  Arms: Default Intervention
Behavioral: Nutrition Education — The nutrition education materials were adapted from materials currently utilized by the Supplemental Nutrition Assistance Education Program
  Arms: Nutrition Education

SUMMARY:
Food insecurity is associated with an increased risk of obesity. The availability of a default option (i.e., option a consumer selects if no active choice is made) has been shown to effectively nudge consumer behavior. An online default option (i.e., prefilled grocery shopping cart) was previously shown to positively impact the food purchases of individuals with food insecurity.The present study aims to extend these findings bye examining efficacy of an online default option in enhancing the nutritional quality of online grocery purchases in individuals with food insecurity over the course of a month.

DETAILED DESCRIPTION:
Food insecurity is associated with an increased risk of obesity and weight-related illnesses. The present study is the first longitudinal randomized control trial to examine if an online prefilled grocery shopping cart (i.e., a default cart) nudges individuals with food insecurity to purchase healthier groceries compared to receiving nutrition education.

It was hypothesized that the prefilled online grocery shopping cart (i.e., default condition) will result in a significant improvement in the nutritional quality of groceries purchased compared to those receiving nutrition education.

Thirty-eight food pantry users recruited from food pantries in New York in 2018 were enrolled in the present study and were given $48.50 to purchase groceries weekly using an online grocery website for five weeks. At baseline, participants were instructed to purchase groceries keeping in mind nutrition, cost, and taste. For the subsequent four weeks (T1-T4), participants were randomized to receive 1) nutrition education or 2) a prefilled online grocery shopping cart that met their nutritional needs based on age and sex (Default).

Our primary nutritional outcomes included HEI scores, calories (kcal), and energy density (kcal/grams).

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Residing in a single person household
3. Receiving assistance at a food pantry
4. Able to read and write in English
5. Able to provide informed consent
6. Current residence in a zip code served by Price Chopper's delivery program
7. None of the following dietary restrictions: Vegetarian/vegan, Gluten-free/celiacs, Lactose intolerance, egg allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Healthy Eating Index Score | 1 month
  (score ranging from 0-100
Calories | 1 month
  kcal
Energy Density | 1 month
  kcal/grams

CONTACTS AND LOCATIONS:
Overall Officials: Julia M Hormes, PhD, Principal Investigator — University at Albany
Locations (1):
- University at Albany, SUNY, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coffino JA, Han GT, Evans EW, Luba R, Hormes JM. A Default Option to Improve Nutrition for Adults With Low Income Using a Prefilled Online Grocery Shopping Cart. J Nutr Educ Behav. 2021 Sep;53(9):759-769. doi: 10.1016/j.jneb.2021.06.011. PMID 34509276